CLINICAL TRIAL: NCT00879346
Title: A Randomised, Open-label, Phase I Study to Determine the Effect of Food on the Pharmacokinetics of Oral AZD8931 Tablets in Healthy Subjects
Brief Title: A Study to Determine the Effect of Food on the Pharmacokinetics of Oral AZD8931 Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Dr Mary Staurt, Medical Science Director, AstraZeneca Pharmaceuticals
Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D0102C00011
Record Dates: First submitted 2009-04-07; First posted 2009-04-10 (Estimated); Last update posted 2009-10-23 (Estimated); Status verified 2009-10

CONDITIONS: Healthy
Keywords: Healthy Volunteers; ADME; Healthy male volunteers
MeSH Terms: interventions — AZD 8931

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): 160mg oral dose of AZD8931
  Interventions: Drug: AZD8931

INTERVENTIONS:
Drug: AZD8931 — 160mg oral single dose (4 x 40mg tablets)

SUMMARY:
Phase I, randomised, open label, 3-period crossover study in healthy male subjects to investigate the effect of food on the pharmacokinetics of AZD8931 and to investigate the safety and tolerability of AZD8931.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Body mass index (BMI) between 19 and 30 kg/m2

Exclusion Criteria:

* Use of any prescribed or non-prescribed medication (including analgesics, herbal remedies, vitamins and minerals) during the two weeks prior to the first administration of investigational product
* Administration of another investigational medicinal product in the 3 months before the start of dosing in this study
* Definite or suspected clinically relevant personal history of adverse drug reactions, or drug hypersensitivity

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2009-03; Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
To investigate the effect of food on the pharmacokinetics of AZD8931 160mg oral dose | Multiple blood PK samples taken between predose to up to 5 days post last dose

SECONDARY OUTCOMES:
To evaluate the safety profile by assessment of adverse events, physical examination, pulse, blood pressure, clinical chemistry, haematology, urinalysis & ECG | Maximus of 7 weeks (From time of consent to last visit including any follow-up)

CONTACTS AND LOCATIONS:
Overall Officials: Emeline Ramos, MD, Principal Investigator — AstraZeneca, Clinical Pharamcology Unit, Alderley Park; Mary Stuart, MD, Study Director — AstraZeneca
Locations (1):
- Research Site, Alderley Park, Cheshire, United Kingdom